CLINICAL TRIAL: NCT06651034
Title: Efficacy of Intralesional Platelet Rich Plasma in Patients of De Quervain's Tenosynovitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mayo-2
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: De Quervain Tenosynovitis
MeSH Terms: conditions — De Quervain Disease

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRP (Experimental): Intralesional Platelet rich plasma
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Other: Platelet Rich Plasma — Under aseptic measures, a phlebotomist obtained the blood in vacutainers. Vacutainers was centrifuged and middle zone containing platelet rich plasma was aspirated in a 5 ml disposable syringe. The patient received intralesional injection

SUMMARY:
De Quervain's tenosynovitis (DQT) was originally identified by Swiss surgeon Fritz de Quervain in 1895. It is a condition involving the entrapment of tendons within the first dorsal compartment of the wrist. In DQT, the sheaths surrounding the abductor pollicis longus (APL) and extensor pollicis brevis tendons thicken as they pass through a fibro-osseous tunnel near the radial styloid of the distal wrist. This thickening leads to pain, which worsens with thumb movements and radial or ulnar deviation of the wrist. Traditional treatment methods, such as corticosteroid injections and physical therapy, often provide only temporary relief and may not address the underlying inflammation effectively. Intralesional platelet rich plasma (PRP) therapy has emerged as a promising alternative, utilizing the patient's own growth factors and cytokines to promote healing and reduce inflammation. By investigating the efficacy of intralesional PRP in patients with DQT, this research aims to provide evidence for a minimally invasive treatment option that could enhance recovery times, reduce pain, and improve functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Either gender,
* Aged between 18 and 60 years
* Presenting with de quervain's tenosynovitis

Exclusion Criteria:

* Previous surgery or intervention forde quervain's tenosynovitis
* Local skin infection or osteomyelitis
* Pregnant or lactating mothers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
VAS Pain Score | 3-week
  The patients were evaluated three weeks after treatment for efficacy. Efficacy was labeled as VAS pain score < 3 after 3 weeks of intralesional PRP injection.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Zarak Awais, MBBS, Principal Investigator — Department of Orthopedic Surgery, Mayo Hospital, Lahore, Pakistan
Locations (1):
- Department of Orthopedic surgery, KEMU/ Affiliated hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No